CLINICAL TRIAL: NCT03340532
Title: HealthSmart: Promoting Healthy Lifestyles for Young Adult Cancer Survivors Using Educational Videos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Prevent Cancer Foundation (Other)
Responsible Party: Principal Investigator, Christopher Recklitis, Ph.D, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-515; R03CA230818-02 (NIH)
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Environmental Exposure to Ultraviolet Light

STUDY DESIGN:
Intervention Model Description: Participants are randomized to view one of two SunSmart educational videos or a control video on sleep hygiene. In the three months following the video intervention, participants' sun protection attitudes and behaviors are assessed. An additional measure of sun protection behaviors 12-months later will be provided by participants who participate in the optional 1-year follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleep hygiene video (Placebo Comparator): Participants will watch a sleep hygiene video
  Interventions: Other: Sleep hygiene video
- Information video (Experimental): The INFORMATION SunSmart video providing basic information about UV risks, including secondary skin cancer and the benefits of SP, as well as specific SP recommendations and steps to integrate SP as part of routine self-care for the healthy cancer survivor
  Interventions: Other: Information SunSmart video
- Information + Appearance video (Experimental): THE INFORMATION + APPEARANCE VIDEO which will include the full information video, along with an additional embedded video segment emphasizing negative appearance consequences of UV exposure.
  Interventions: Other: THE INFORMATION + APPEARANCE VIDEO

INTERVENTIONS:
Other: THE INFORMATION + APPEARANCE VIDEO — THE INFORMATION + APPEARANCE VIDEO which will include the full information video, along with an additional embedded video segment emphasizing negative appearance consequences of UV exposure.
  Arms: Information + Appearance video
Other: Information SunSmart video — The INFORMATION SunSmart video providing basic information about UV risks, including secondary skin cancer and the benefits of SP, as well as specific SP recommendations and steps to integrate SP as part of routine self-care for the healthy cancer survivor
  Arms: Information video
Other: Sleep hygiene video — Contain information on better sleep hygiene
  Arms: Sleep hygiene video

SUMMARY:
To assess the efficacy of the two SunSmart intervention videos to change sun protection attitudes and behaviors

DETAILED DESCRIPTION:
SunSmart is a novel video intervention designed to prevent secondary skin cancer in young adult cancer survivors by increasing their adherence to recommended sun protection.

This study will assess two versions of the SunSmart video intervention. These are: 1) The INFORMATION VIDEO providing basic information about UV risks, including secondary skin cancer and the benefits of sun protection (SP), as well as specific SP recommendations and steps to integrate SP as part of routine self-care for the healthy cancer survivor; and 2) THE INFORMATION + APPEARANCE VIDEO which will include the full information video, along with an additional embedded video segment emphasizing negative appearance consequences of UV exposure. Primary aim of the study is to assess the impact of the video intervention on sun protection intentions and behavior in young adult cancer survivors compared to a control intervention. Secondary aims are to describe the impact of the appearance information when included in the SunSmart intervention, to investigate the extent to which the intervention changes sun protection through hypothesized mediating variables, and to describe the consistency of sleep behaviors over time in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* History of cancer diagnosis at least one year prior
* Current age 18-35
* No cancer therapy in the prior 3 months (excluding chemoprevention agents)
* No future cancer therapy planned
* Able to read and write in English
* Not compliant with recommended sun protection, as determined by at least one of the following criteria:

  1. Any intentional sunbathing, artificial tanning or a sunburn in the past 5 years; OR
  2. Having a moderate to light complexion (Fitzpatrick skin types I-IV), and not using sunscreen ≥ 90% of the time during incidental sun exposure.

Exclusion Criteria:

* History of skin cancer diagnosis
* Enrolled on DFCI protocol 17-385 or any other sun protection intervention in the past 5 years.
* Any impairment (e.g., hearing, visual, cognitive) that interferes with the ability to complete all measures independently

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-09-28 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Change in SP Index scores from baseline to post-summer assessment | 3 months
  SP index is comprised of 15 self-report items assessing SP Behaviors

SECONDARY OUTCOMES:
Perceived appearance vulnerability | one month
  2 items assessing perceived likelihood that UV exposure will lead to negative appearance changes
Perceived health and appearance benefit | one month
  8 self-report items assessing expected benefits to SP
Perceived health vulnerability | one month
  2 items assessing perceived likelihood that UV exposure will lead to future skin cancers.
SP Intentions | one month
  13 items measuring intentions to practice SP
Insomnia symptoms | one month
  7 -item Insomnia Severity Scale (ISS). Total ISS scale scores range from a low of 0 (least insomnia) to a high of 28 (worst insomnia)
Change in SP Index scores from post-summer assessment to one year later | 12-months
  SP index is comprised of 15 self-report items assessing SP Behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Recklitis, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No